CLINICAL TRIAL: NCT00175864
Title: Open Label, Multicenter Study of the Safety and Efficacy of Oral Treatment With Immediate Release Seletracetam (Ucb 44212) at Individualized Doses up to a Maximum of 160mg/Day in Refractory Epileptic Patients.
Brief Title: Open Label Study (Everyone Who Participates Receives Drug) to Further Determine How Safe and Effective Oral Treatment of Seletracetam is in Patients With Refractory Epilepsy.
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01212; Not yet available
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Epilepsy
Keywords: Partial Onset, Primary Generalized Seizures, Seletracetam
MeSH Terms: conditions — Epilepsy | interventions — Seletracetam

INTERVENTIONS:
Drug: Seletracetam (ucb 44212)

SUMMARY:
This is a safety and efficacy study of add on therapy with seletracetam in patients experiencing refractory epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* An IRB/IEC approved written informed consent form signed and dated Male/Female patients age 18 (or 16 years where permitted by law) to 65.
* Minimum body weight of 40 kg.
* Patients with a confirmed diagnosis of refractory epilepsy of ≥ 6 months.
* Patients must be receiving 1 - 3 concomitant AEDs.
* Female patients without childbearing potentials (2 years post-menopausal or surgical sterilization) are eligible. Female patients with childbearing potential are eligible if they use a medically accepted non-hormonal contraceptive method.

Exclusion Criteria:

* Seizures occurring in clusters (seizures occurring either too frequently or indistinctly separated to be reliably counted).
* Status epilepticus within 3 months of Visit 1.
* History of non-epileptic seizures.
* Patients on vigabatrin.
* Patients on felbamate, unless treatment has been continuous for ≥ 18 months.
* Use of benzodiazepines (for any indication) taken at a higher frequency than an average of once a week, unless counted as one of the concomitant AEDs.
* Ongoing psychiatric disease other than mild controlled disorders.
* Patients with a clinically significant organ dysfunction.
* Known allergic reaction or intolerance to pyrrolidine derivatives and/or excipients.
* Pregnant or lactating women. Any woman with childbearing potential who is not using a medically accepted, non-hormonal method of birth control.

Ages: 16 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-02

PRIMARY OUTCOMES:
Safety profile of seletracetam

SECONDARY OUTCOMES:
Reduction in seizure frequency

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Bennett, PhD, Study Director — UCB Pharma